CLINICAL TRIAL: NCT05121532
Title: Evaluation of Serum Interleukin-15 and Interleukin-22 Levels in Patients With Non-segmental Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Samah Saeed Badrous, resident doctor at dermatology department balina central hospital, Sohag University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-21-11-12
Record Dates: First submitted 2021-11-14; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non segmental vitiligo (Active Comparator): serum analysis
  Interventions: Diagnostic Test: Interleukin-15 and Interleukin-22
- normal volunteer (Active Comparator): serum analysis
  Interventions: Diagnostic Test: Interleukin-15 and Interleukin-22

INTERVENTIONS:
Diagnostic Test: Interleukin-15 and Interleukin-22 — Serum Interleukin-15 and Interleukin-22 in non segmental vitiligo

SUMMARY:
Evaluation of Serum Interleukin-15 and Interleukin-22 Levels in Patients with Non-segmental Vitiligo before and after phototherapy

DETAILED DESCRIPTION:
This prospective study will include 30 patients with NSV, attending the Outpatient Clinics of Dermatology at Sohag University Hospitals, as well as 30 normal volunteers as control.

This study will be submitted for approval by Research and Ethical committees at Sohag Faculty of Medicine. An informed written consent will be obtained from each subject prior to participation in the study after full explanation of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* • Patients suffering from non segmental vitiligo.

  * Patients not on medical treatment or phototherapy for vitiligo in the last 3 months.

Exclusion Criteria:

* • Patients with systemic or cutaneous inflammatory disorders.

  * Patients on treatment for vitiligo in last 3 months.
  * Pregnant and lactating patients.
  * Patients with history of diabetes.
  * Patients with history of autoimmune diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Serum Interleukin-15 and Interleukin-22 Levels | 3 months
  3 ml venous blood will be obtained from participante using commerciall available double antibody sandwich enzyme-linked immunosorbent assay (ELISA) kits to evaluate
  1. Serum IL15 level .
  2. Serum IL22 level. 3 ml venous blood will be obtained from participante using commerciall available double antibody sandwich enzyme-linked immunosorbent assay (ELISA) kits to evaluate
  1. Serum IL15 level . 2. Serum IL22 level.